CLINICAL TRIAL: NCT04336072
Title: Trial of Reminder Focused Positive Psychiatry in Comorbid Attention Deficit Hyperactive Disorder With Posttraumatic Stress Disorder
Brief Title: Reminder Focused Positive Psychiatry in Adolescents With ADHD and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Kern Medical (Unknown); American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Principal Investigator, Naser Ahmadi, MD, PhD, Assistant Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # 16030
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Posttraumatic Stress Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent from parents and informed assent from eligible adolescents with comorbid ADHD and PTSD, participants will be randomized into: a) RFPP group therapy or trauma focused cognitive behavioral group therapy
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomly assigned to groups. Outcome assessors will be blinded to participants and interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminder Focused Positive Psychiatry (RFPP) (Experimental): RFPP aims to enhance contextual discrimination and emotional regulation, and promote the use of adaptive coping strategies in response to trauma reminders, including recognizing reminders, shifting attention from intrusive memories during exposure to reminders to a focus on positive feelings, thoughts, goals, and choices
  Interventions: Behavioral: RFPP
- Trauma Focused Cognitive Behavioral Therapy (TFCBT) (Active Comparator): TFCBT is inclusive of the trauma narrative (TN) & processing components facilitated the child talking about memories individually and in groups, the last sessions focused on grief-specific elements.
  Interventions: Behavioral: TFCBT

INTERVENTIONS:
Behavioral: RFPP
  Arms: Reminder Focused Positive Psychiatry (RFPP)
Behavioral: TFCBT
  Arms: Trauma Focused Cognitive Behavioral Therapy (TFCBT)

SUMMARY:
This feasibility study investigates the impact of reminder-focused-positive-psychiatry (RFPP) on attention-deficit-hyperactive-disorder (ADHD) and posttraumatic-stress-disorder (PTSD) symptoms, vascular-function, inflammation and well-being of adolescents with comorbid ADHD & PTSD.

In this randomized clinical trial, 24 subjects with comorbid ADHD and PTSD, aged 12-18 years old, free of known medical and other major psychiatric disorders, will be recruited from the pool of eligible subjects at Los Angeles and Kern County Children Mental Health Centers (>1500 subjects) after obtaining informed consent from parents as well as subjects' assentment. Commonwealth and Oswell Kern County Mental Health Clinic will be used for subjects enrollment, randomization as well as study implementation from trauma disorder clinic. Kern Medical will be used for manuscript write up and analyses.

Adolescents will be randomized to: group-RFPP or trauma-focused group-cognitive-behavioral-therapy (TF-CBT). Participants will complete twice-weekly-intervention for 6-weeks-trial. The group-RFPP-intervention will be inclusive of RFPP interventions on a) traumatic-reminders, and b Avoidance & negative-cognition. Vascular-function-measured as temperature-rebound (TR), C-reactive-protein (CRP), homocysteine, SNAP-questionnaire, Clinician-Administered PTSD-Scale-children-version (CAPS-CA) and neuropsychiatric-measures will be measured at baseline and 6th week. Subjects will be followed for 12 months.

Parents and subjects will be informed of the risks associated with use of venipuncture and loss of confidentiality of collected information.

DETAILED DESCRIPTION:
PTSD and ADHD are major public health problems. Many individuals with comorbid ADHD and PTSD continue to suffer despite treatment with FDA approved medications including antidepressants (sertraline and paroxetine), prazosin and/or the Institute of Medicine approved psychotherapy. Long-term outcomes with even the most intensive treatments, although significant, were modest, and reveal persistent morbidity and disability for many individuals with PTSD, especially in those with comorbid ADHD.19 While current treatments focused on treatment to reduce the associated suffering and disability of morbid ADHD and PTSD. These interventions are, however, not sufficient to promote human welfare, improve levels of positive psychosocial characteristics (PPCs), and resilience. Positive psychiatry (PP) focuses on promoting well-being, enhancing behavioral and mental wellness in both youth and adults20, however its impact on youth with comorbid PTSD and ADHD has not been studied. We hypothesize that PP intervention would significantly enhance vascular function, resilience, wellbeing, increase posttraumatic growth and reduce inflammation in morbid ADHD and PTSD. This randomized trial will the first to investigate the impact of psychiatric positive interventions, as opposed to intervention on ameliorating vulnerability, on adolescents with morbid ADHD and PTSD. Findings of this study can provide a better understanding of impact of PP on psychiatric and biomolecular characteristics of adolescent with PTSD and ADHD. If successful, this proposal will be available for large scale studies following which it could potentially be deployed in daily clinical practice.

RESEARCH METHOD:

In this randomized clinical trial, the three related and overlapping specific aims are directed to examine the feasibility of PP intervention, as well as its impact on positive psychological wellbeing, and neurovascular inflammation in adolescent subjects with comorbid ADHD and PTSD.

Synopsis. In this randomized clinical trial, 24 subjects with comorbid ADHD and PTSD, aged 12-18 years old, free of known medical and other major psychiatric disorders, will be recruited from the pool of eligible subjects at Los Angeles and Kern County Children Mental Health Centers (>1500 subjects) after obtaining informed consent from parents as well as subjects' assentment. Commonwealth and Oswell Kern County Mental Health Clinic will be used for subjects enrollment, randomization as well as study implementation from trauma disorder clinic. Kern Medical will be used for manuscript write up and analyses.

Parents and subjects will be informed of the risks associated with use of venipuncture and loss of confidentiality of collected information. Eligible subjects will be randomized to 1) PP group intervention, or 2) control condition group (12 in each group) for 6 week intervention and 6 week of follow up.

Recruited subject will be followed before, during and after interventions. Both groups will be on adequate stimulant therapy for ADHD. Group PP intervention consists of 12 sessions of group PP in 6 week that will be completed by the participant with the guidance of a trainer. Sham control condition consists of 12 sessions in 6 week of group exercises that will be completed by the participant with the guidance of a trainer.

All subjects will undergo radial artery flow mediated dilatation, a measure of vascular function, venipuncture for measuring of CRP, homocysteine and IL-6, as well as completion of positive psychiatry and wellbeing batteries at baseline, 3rd and 6th of intervention and 12th week follow up.

A- Measurements A1.History and Physical Exam (H&P): All consented patients will undergo a baseline H&P, intervention, and post-trial observation periods by a physician.

A2. Medications: All medications during pre-trial, intervention and post-trial will be charted A3. Psychiatry Batteries: SNAP teacher and parent questionnaire, Positive Psychotherapy Inventory, VIA Survey of Character Strengths, PERMA, PANAS, optimism, posttraumatic growth inventory, Connor Davidson resilience scale, Clinician Administered PTSD Scale (CAPS) children version will be measured at baseline, 3rd, 6th and 12th week.

A4. Vascular Function Assessment via FMD: After resting in a supine position in a room with temperature 23° to 25° C for 30 minutes, brachial artery endothelial function will be assessed noninvasively by ultrasound using reactive hyperemia procedure. Brachial artery diameter above antecubital crease will be measured at least 60 cycles from baseline to 5 min cuff inflation, and 5 min post cuff deflation.

A5.Venipuncture and laboratory measurements: Venous blood samples of all subjects after 8 hours of fasting will be drawn at baseline, 3rd, 6th and 12th week. The assessment of C-reactive protein (CRP) and homocysteine will be performed using the standard techniques. The concentrations of IL-6 will be determined using commercially available solid-phase sandwich enzyme-linked immunosorbent assay kits. The range of detection is 15-1540 pg/ml for IL-6.21

B- Interventions:

B1.Reminder Focused Positive Psychiatry: RFPP group will receive 6 week (12 sessions and 12 exercises) of positive psychiatry to improve wellbeing. The group PP exercises are inclusive of Posttraumatic Growth, Resilience, Gratitude and Optimism, Self-regulation and Personal Strength, Enjoyable and meaningful activities, Personal mastery and self-efficiency. Groups last approximately 60 minutes, and positive responding (responding to others in an active and constructive way), personal strengths, gratitude, forgiveness and identifying positives from negative situations will be included. Nondirective prompts will be used to stimulate in-depth discussion. Feedback from subjects will be captured. All facilitators have experience of facilitating therapeutic groups and of working with individuals with a diagnosis of ADHD and PTSD. Facilitators participate in all exercises themselves, they share personal examples from their own lives with the group, and are encouraged to do the 'ongoing exercise' in their own time. Participants are not prohibited from sharing distressing, unpleasant, or negative states and experiences in the group. Negative contributions are validated but not focused on. Instead, facilitators establish a link between the negative experience and one or more of the intervention's target areas.

C. Statistical Analysis:

All statistical analyses will be performed during the last 4 months of the study. T test and Chi Square test will be used to assess differences between groups. The association between PP and control condition will be analyzed by linear and mixed regression analyses. In addition, the change in overall symptoms, ADHD and PTSD specific symptoms, and neurovascular inflammation in response to PP will be evaluated. These analyses will be adjusted for demographics, mental and medical covariates.

D. Sample Size for Specific Aim 1-3:

A measurable change in vascular function and increase in PERMA are outcomes of interest. The sample size of 12 per group that has been chosen based on priori study, will detect a 20% difference in vascular function and PERMA score amongst groups, with a study power of 0.8 and significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* English speaking Boy/Girl Age 9 - 18 years old
* Able to read/write in English
* Documented ADHD and PTSD, and parents provided informed consent

Exclusion Criteria:

* Psychotic or Mood Disorders or Self-injurious behavior
* Cognitive disorder or other neurodevelopmental disorders
* Diagnosis of substance use disorder

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Acceptability of RFPP to treat adolescents with PTSD and ADHD | 12 month
  Measure the acceptability after 6-week intervention where both adolescents and parents will be asked about overall satisfaction with treatment using the validated and reliable Client Satisfaction Questionnaire (CSQ-8).
  The aim is a mean above 20.00 (Good-Excellent) on the 8 to 32 scale of CSQ-8, and sessions' mean of 4.00 (very valuable session) on the 0 to 5 Session Feedback Questionnaire scale (SFQ).
Feasibility of RFPP to treat adolescents with PTSD and ADHD | 12 month
  Measure the feasibility of RFPP intervention measured by retention rate of participants in RFPP group post-intervention.
  The goal is a ≥50% referred-to-enrolled rate, ≥70% intervention completion rate and 70% 12-month follow up.
Fidelity of RFPP to treat adolescents with PTSD and ADHD | 12 month
  Measure the adherence and competence of therapists to the model will be assessed by live observation, role play and provider self-report and checklist. Session will observed or listened to as they are happening. Therapists demonstrate specific skills which might use with a client generically and as applied to specific clinical cases required by the model. Therapists describe in detail exactly what they do in the session and how the client respond, also complete checklists following sessions.
  Interrater reliability will be assessed using the chance-corrected weighted kappa statistic from 0-1, with aim of 0.8+ (almost perfect agreement).

SECONDARY OUTCOMES:
Change in PTSD symptoms in response of RFPP at 6-week intervention and 12-month follow up. | 12 month
  Measure the change in reactivity of trauma reminder and core PTSD symptoms in response to RFPP at 6-week intervention and 12-month follow up, compared to changes in such measures in response to TFCBT.
  The change in reactivity to trauma reminder - assessed with UCLA Trauma Reminder Inventory questionnaire with range of 0 to 88- , PTSD core symptoms - assessed by Clinician Administered PTSD Scale children version (CAPS-CA) questionnaire with range of 0 to 160. All measures demonstrated acceptable internal consistency.
Change in ADHD symptoms in response of RFPP at 6-week intervention and 12-month follow up. | 12 month
  Measure the change in core ADHD symptoms in response to RFPP at 6-week intervention and 12-month follow up, compared to changes in such measures in response to TFCBT.
Change in mental wellbeing in response of RFPP at 6-week intervention and 12-month follow up. | 12 month
  Measure the change in positive biopsychosocial trait, mental wellbeing and parent-child interactions in response to RFPP at 6-week intervention and 12-month follow up, compared to changes in such measures in response to TFCBT.
  The percent of change in questionnaires of PERMA (Positive emotion, engagement, relationships, meaning, and accomplishment), gratitude, posttraumatic growth inventory, Connor-Davidson resilience scale, and PACHIQ (Parent-Child Interaction Questionnaire) with range of 0- 100%, where 60%+ represent optimal biopsychosocial trait and wellbeing. All measures demonstrated acceptable internal consistency.
Change in physiologic biomarkers in response of RFPP at 6-week intervention and 12-month follow up. | 12 month
  Measure the change in fingertip vascular function, C reactive protein (CRP) and homocysteine in response to RFPP at 6-week intervention and 12-month follow up, compared to changes in such measures in response to TFCBT.
  The change in digital thermal monitoring (DTM) of fingertip vascular function - through reactive hyperemia procedure, range ratio of -1 to 2.5 - CRP with range of 0-50 mg/L, and homocysteine with range of 0-100 mcmol/L. All measures are standardized and demonstrated acceptable internal consistency.
Change in the rate of psychiatric hospitalization and suicidality in response of RFPP at 6-week intervention and 12-month follow up. | 12 month
  Measure the change in rate of psychiatry hospitalization and suicidality in response to RFPP at 6-week intervention and 12-month follow up, compared to changes in such measures in response to TFCBT.
  The percent change in the rate of psychiatry hospitalization and suicidality, number and frequency of such events. All verified by clinicians blinded to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Naser Ahmadi, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Kern, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmadi N, Chaudhry S, Salam T, Rodriguez J, Kase M, Olango G, Molla M, McCracken J, Pynoos R. A Randomized Controlled Feasibility Trial of Reminder-Focused Positive Psychiatry in Adolescents With Comorbid Attention-Deficit/Hyperactivity Disorder and Posttraumatic Stress Disorder. Prim Care Companion CNS Disord. 2020 Sep 3;22(5):19m02579. doi: 10.4088/PCC.19m02579. PMID 32898346